CLINICAL TRIAL: NCT03395067
Title: Multidisciplinary Treatment of Obesity Prior to In Vitro Fertilization: Impact on Global Reproductive Outcomes
Brief Title: Multidisciplinary Treatment of Obesity Prior to in Vitro Fertilization: Impact on Global Reproductive Outcomes (PRO-FIV Study)
Acronym: PRO-FIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Gemma Casals i Soler, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCB/2017/0730
Record Dates: First submitted 2017-12-17; First posted 2018-01-10 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Obesity; Infertility
Keywords: Obesity; Infertility; In vitro fertilization
MeSH Terms: conditions — Obesity; Infertility

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial including 2 arms: intervention group and control group.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle counseling (Active Comparator)
  Interventions: Behavioral: Intervention group
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Intervention group — Lifestyle counseling coupled with psychotherapeutical intervention
  Arms: Lifestyle counseling

SUMMARY:
The aim of the present study is to evaluate the impact of a multidisciplinary treatment of obesity prior to IVF on global reproductive outcomes and maternofetal metabolic and cardiovascular risk factors.

This is a randomized controlled trial in obese infertile women before starting an IVF cycle. The intervention is based on a structured multidisciplinary program in support groups, which includes diet, physical activity and psychological therapy. IVF will be started immediately after this therapy. Patients included in the control group will start an IVF cycle immediately after the randomization. The results of this study may allow the identification of patients who would benefit from obesity treatment, so as to establish appropriate preventive and therapeutic strategies and to reduce the maternal obesity impact in future generations.

DETAILED DESCRIPTION:
The aim of the present study is to evaluate the impact of a multidisciplinary treatment of obesity prior to IVF on global reproductive outcomes and maternofetal metabolic and cardiovascular risk factors.

This is a randomized controlled trial in obese infertile women (body mass index ≥30 kg/m2) before starting an IVF cycle. In the intervention group, the aim is a weight loss of at least 10% in a 16-week period of treatment based on a multidisciplinary approach and support groups, which includes diet, physical activity and psychological therapy. IVF will be started immediately after this period. Patients included in the control group will start an IVF cycle immediately after the randomization. The results of this study may allow the identification of patients who would benefit from obesity treatment, so as to establish appropriate preventive and therapeutic strategies and to reduce the maternal obesity impact in future generations.

ELIGIBILITY:
Inclusion Criteria:

* Obese infertile patients (body mass index ≥ 30 Kg/m2) prior to an in vitro fertilization cycle

Exclusion Criteria:

* Pathological conditions: diabetes type I, Cushing syndrome, premature ovarian failure, uncontrolled thyroidal dysfunction, hepatic and/or renal dysfunction, antiphospholipid syndrome, medical condition that contraindicate ovarian stimulation and/or pregnancy
* Simultaneous practice of another strategy to lose weight
* Physical conditions limiting exercise training
* Patients unable to understand spanish language or to give informed consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2018-01-28 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
live birth rate of a healthy baby in a non-complicated pregnancy | 10 months after starting the IVF treatment
  live birth rate in a pregnancy without major complications: gestational diabetes, hypertensive disorders, preterm delivery, congenital anomalies, stillbirth, neonatal death, shoulder dystocia, maternal venous thromboembolism, fetal growth abnormal outcomes (macrosomia, large for gestational age, intrauterine growth restriction)

SECONDARY OUTCOMES:
anthropometric parameters: weight (kilograms) | 4 months after starting the intervention
  weight change during intervention, measured in kilograms
anthropometric parameters: body mass index - BMI (kilograms/metro2) | 4 months after starting the intervention
  BMI change during intervention, measured as kilograms/metro2
anthropometric parameters: abdominal circumference (centimeters) | 4 months after starting the intervention
  abdominal circumference change during intervention measured in centimeters
hormonal parameters: antimullerian hormone (AMH) | 2 years (simultaneous analysis of all the biological samples)
  AMH serum levels before the intervention (intervention group) and before the IVF (2 arms)
hormonal parameters: insulin | 2 years (simultaneous analysis of all the biological samples)
  insulin serum levels before the intervention (intervention group) and before the IVF (2 arms)
hormonal parameters: leptin | 2 years (simultaneous analysis of all the biological samples)
  leptin serum levels before the intervention (intervention group) and before the IVF (2 arms)
hormonal parameters: adiponectin | 2 years (simultaneous analysis of all the biological samples)
  adiponectin serum levels before the intervention (intervention group) and before the IVF (2 arms)
hormonal parameters: ghrelin | 2 years (simultaneous analysis of all the biological samples)
  ghrelin serum levels before the intervention (intervention group) and before the IVF (2 arms)
IVF outcomes: cycle cancellation rate | 3 months after starting IVF cycle
  cycle cancellation rate: cancelled cycles/ initiated cycles
IVF outcomes: gonadotropin doses (UI) | 3 months after starting IVF cycle
  total gonadotropin doses used in the IVF stimulation protocol
IVF outcomes: number of oocytes | 3 months after starting IVF cycle
  number of oocytes retrieved
IVF outcomes: number of embryos | 3 months after starting IVF cycle
  total number of embryos obtained in 2 pronuclear stage
IVF outcomes: number of good quality embryos | 3 months after starting IVF cycle
  number of good quality embryos (type A and B) obtained in the cleavage stage
IVF outcomes: clinical pregnancy rate | 3 months after starting IVF cycle
  clinical pregnancy rate: clinical pregnancies/started cycles
IVF outcomes: miscarriage rate | 3 months after starting IVF cycle
  miscarriage rate: miscarriages/clinical pregnancies
fetal ultrasound | 26-30 weeks after confirmation of pregnancy
  fetal ultrasound and Doppler parameters at 28-32 weeks of gestation. All parameters are measured according to the current guidelines and reported as quantitative measurements.
postpartum anthropometric outcomes: maternal abdominal circumference (centimeters) | 12 months after the delivery
  Maternal abdominal circumference in centimeters 1 month and 12 months after the delivery
postpartum anthropometric outcomes: maternal weight (kilograms) | 12 months after the delivery
  Maternal weight in kilograms 1 month and 12 months after the delivery
postpartum anthropometric outcomes: neonatal weight (grams) | 12 months after the delivery
  neonatal weight in grams 1 month and 12 months after the delivery
postpartum anthropometric outcomes: neonatal height (centimeters) | 12 months after the delivery
  neonatal height in centimeters 1 month and 12 months after the delivery
postpartum anthropometric outcomes: neonatal skin fold measurements (millimeters) | 12 months after the delivery
  neonatal skin fold measurements in millimeters 1 month and 12 months after the delivery

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Casals, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain